CLINICAL TRIAL: NCT07401693
Title: The Effect of Oral Health Care Program on Oral Hygiene and Oral Function for the Elderly Patient With Dementia in Day Care Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiou-fang Lu (Other)
Responsible Party: Sponsor-Investigator, Shiou-fang Lu, Assistant Professor, Tzu Chi University
Organization: Tzu Chi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB23-01-003
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dementia; Oral Health Care; Oral Hygiene
Keywords: Dementia; Oral hygiene; Day care center; Older adults; oral care intervention; oral function
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either an intervention group or a control (waiting-list) group. The intervention group received the oral health care program, while the control group did not receive the intervention during the study period. Outcomes were assessed at baseline and at 4 weeks after the intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Outcome assessors were blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Health Care Program (Experimental): Participants assigned to the intervention group received a structured oral health care program designed to improve oral hygiene and oral function. Outcome measures were assessed at baseline and at 4 weeks after the intervention.
  Interventions: Behavioral: Oral Health Care Program
- Usual Care (Waiting-list Control) (No Intervention): Participants assigned to the control (waiting-list) group did not receive the oral health care intervention during the study period and continued with usual care. Outcome measures were assessed at baseline and at 4 weeks.

INTERVENTIONS:
Behavioral: Oral Health Care Program — A structured oral health care program designed to improve oral hygiene and oral function among older adults with dementia attending a day care center. The program included guided oral exercises and daily oral hygiene practices delivered over a 4-week period.
  Arms: Oral Health Care Program

SUMMARY:
This study evaluated the effects of an oral health care program on oral hygiene and oral function in older adults with dementia attending a day care center. Participants received a structured oral health care intervention, and changes in oral hygiene and oral function were assessed over a 4-week follow-up period. The goal of this study was to explore whether a structured oral health care program could help improve oral health outcomes in older adults with dementia in a day care setting.

DETAILED DESCRIPTION:
This study employed a quasi-experimental design to examine the effects of an oral health care program on oral hygiene and oral function among older adults with dementia attending a day care center. Participants received a structured oral health care intervention designed to promote oral hygiene practices and oral functional ability. Outcome measures related to oral hygiene and oral function were assessed at baseline and at 4 weeks after the intervention. This study aimed to provide evidence on the effectiveness of an oral health care program for improving oral health outcomes in older adults with dementia in a day care setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 60 years or older.
2. Diagnosed with dementia by a physician.
3. Attending a day care center.
4. Able to participate in the oral health care program and assessments.
5. Provided informed consent from the participant or a legally authorized representative

Exclusion Criteria:

1. Presence of acute medical conditions that would interfere with participation.
2. Severe physical or mental conditions that prevent completion of the intervention or outcome assessments.
3. Refusal or inability to provide informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Oral hygiene | From baseline to 4 weeks after intervention
  Oral hygiene was assessed using the Oral Health Assessment Tool (OHAT) as the primary outcome measure. OHAT is a validated composite scale with a total score ranging from 0 to 16, with higher total scores indicating poorer oral health status.
Oral function | From baseline to 4 weeks after intervention
  Oral function was assessed using standardized functional assessments to evaluate changes in oral motor and swallowing function following the oral care intervention. Higher scores or values indicate better oral or swallowing function.

SECONDARY OUTCOMES:
Plaque index | From baseline to 4 weeks after intervention
  Dental plaque accumulation was assessed using the Plaque Index, which evaluates the thickness of dental plaque at the gingival area. Scores range from 0 to 3, with higher scores indicating greater plaque accumulation and poorer oral hygiene.
Tongue coating index | From baseline to 4 weeks after intervention.
  Tongue coating was assessed using the Tongue Coating Index, with scores ranging from 0 to 2. A lower score indicates less tongue coating and better oral hygiene.
Puff cheeks | From baseline to 4 weeks after intervention.
  The ability to puff the cheeks was assessed using a functional scoring scale ranging from 0 to 5, where 0 indicates inability to puff the cheeks, 3 indicates barely able to puff the cheeks, and 5 indicates the ability to puff both cheeks. Higher scores indicate better oral function.
Choke | From baseline to 4 weeks after intervention.
  Swallowing ability was assessed using a choking frequency scale ranging from 0 to 5, where 0 indicates tube feeding, 1 indicates frequent choking, 3 indicates occasional choking, and 5 indicates almost no choking. Higher scores indicate better swallowing function.
Repetitive Saliva Swallowing Test (RSST) | From baseline to 4 weeks after intervention.
  Have the subject sit. The examiner gently places their fingertip on the subject's Adam's apple or hyoid bone and instructs the subject to swallow saliva. The examiner can feel the Adam's apple rise and then return to its original position. If the subject experiences dry mouth, about 1 cc of water can be given. Observe this action for 30 seconds and record the number of swallows obtained through palpation.The Repetitive Saliva Swallowing Test (RSST) was used to assess swallowing function by counting the number of saliva swallows within 30 seconds. Higher values indicate better swallowing ability.
Oral DDK rate(times/10') | From baseline to 4 weeks after intervention.
  Oral diadochokinetic (DDK) rate was assessed by counting the number of syllable repetitions produced within 10 seconds. Higher values indicate better oral motor function.

CONTACTS AND LOCATIONS:
Locations (1):
- Mennonite Christian Hospital Shoufeng Branch Day Care Center, Hualien City, Hualien County, Taiwan

IPD SHARING:
Plan to Share IPD: No